CLINICAL TRIAL: NCT05608291
Title: A Phase 3 Trial of Fianlimab (Anti-LAG-3) and Cemiplimab Versus Pembrolizumab in the Adjuvant Setting in Patients With Completely Resected High-risk Melanoma
Brief Title: A Trial to See if the Combination of Fianlimab With Cemiplimab Works Better Than Pembrolizumab for Preventing or Delaying Melanoma From Coming Back After it Has Been Removed With Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3767-ONC-2055; 2022-501576-25-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2022-10-14; First posted 2022-11-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Melanoma
Keywords: Resected High Risk Melanoma; Skin Cancer; Stage IIB; Stage IIC; Stage III; Stage IV; LAG-3 Lymphocyte activation gene 3; Adjuvant Setting; anti-PD-1 Monoclonal Antibody
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — cemiplimab; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fianlimab HD + Cemiplimab (Experimental): Patients will be administered one combination dose of fianlimab high dose (HD) and cemiplimab
  Interventions: Drug: Fianlimab; Drug: Cemiplimab
- Fianlimab LD + Cemiplimab (Experimental): Patients will be administered one combination dose of fianlimab low dose (LD) and cemiplimab
  Interventions: Drug: Fianlimab; Drug: Cemiplimab
- Pembrolizumab (Active Comparator): Patients will be administered one dose of pembrolizumab co-infused with saline/dextrose placebo
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Fianlimab — Fianlimab will be administered by intravenous (IV) infusion every (Q) 3 weeks
  Other Names: REGN3767
  Arms: Fianlimab HD + Cemiplimab; Fianlimab LD + Cemiplimab
Drug: Cemiplimab — Cemiplimab will be administered by IV infusion Q 3 weeks
  Other Names: REGN2810; Libtayo
  Arms: Fianlimab HD + Cemiplimab; Fianlimab LD + Cemiplimab
Drug: Pembrolizumab — Pembrolizumab will be administered by IV infusion Q 3 weeks
  Other Names: MK-3475; lambrolizumab; Keytruda
  Arms: Pembrolizumab
Drug: Placebo — Matching placebo co-infused with pembrolizumab IV, will be administered by IV infusion Q 3 weeks
  Arms: Pembrolizumab

SUMMARY:
This study is researching an experimental drug called REGN3767, also known as fianlimab (R3767), when combined with another medication called cemiplimab (each individually called a "study drug" or called "study drugs" when combined) compared with an approved medication called pembrolizumab.

The objective of this study is to see if the combination of fianlimab and cemiplimab is an effective treatment compared to pembrolizumab in patients that have had melanoma removal surgery but are still at high risk for the recurrence of the disease. Pembrolizumab is an approved treatment in some countries in this clinical setting.

The study is looking at several other research questions, including:

* What side effects may happen from receiving the study drugs.
* How much study drug is in the blood at different times.
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects). Antibodies are proteins that are naturally found in the blood stream that fight infections.
* How administering the study drugs might improve quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

1. All patients must be either stage IIB, IIC, III, or stage IV per American Joint Committee on Cancer (AJCC) 8th edition and have histologically confirmed melanoma that is completely surgically resected in order to be eligible as defined by the protocol
2. Complete surgical resection must be performed within 12 weeks prior to randomization, and enrollment may occur only after satisfactory wound healing from the surgery
3. All patients must have disease-free status documented by a complete physical examination and imaging studies within 4 weeks prior to randomization, as described in the protocol

Key Exclusion Criteria:

1. Uveal melanoma
2. Any evidence of residual disease after surgery by imaging, pathology, or cytology.
3. Ongoing or recent (within 2 years) evidence of clinically significant autoimmune disease that required treatment
4. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C (HCV) infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection, as described in the protocol
5. Another malignancy that is currently progressing or that required active treatment in the past 5 years, as described in the protocol
6. Participants with a history of myocarditis
7. Adolescent patients (≥12 to <18 years old) with body weight <40 kg

Note: Other Protocol Defined Inclusion/ Exclusion Criteria Apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1564 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2028-05-16 (Estimated); Study Completion 2030-02-15 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival (RSF) | Up to 5 Years
  Time from randomization to the first documented recurrence of disease at any site (excluding new primary melanomas) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Distant metastasis-free survival (DMFS) | Up to 5 Years
  Time between the date of randomization and the date of the first distant metastasis.
Overall survival (OS) | Up to 5 Years
  Time from randomization to the date of death.
Occurrence of treatment-emergent adverse events (TEAEs) | Up to 5 Years
  A TEAE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Occurrence of immune-mediated EAEs (im-EAEs) | Up to 5 Years
  imAEs are a unique set of toxicities thought to be caused by unrestrained cellular immune responses.
Occurrence of serious adverse events (SAEs) | Up to 5 Years
  An SAE is any untoward medical occurrence that at any dose:
  * Results in death - includes all deaths, even those that appear to be completely unrelated to study drug (eg, a car accident in which a patient is a passenger).
  * Is life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect.
  * Is an important medical event
Occurrence of adverse events of special interest (AESIs) | Up to 5 Years
  An AESI (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it
Occurrence of TEAEs resulting in death | Up to 5 Years
  A TEAE resulting in death is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Occurrence of dose-limiting toxicity (DLT) | Up to 5 Years
  A DLT is defined as a study-drug related TEAE, including imAEs, that could preclude enrolling additional adolescent patients at the selected dose. Dose-limiting toxicity will be evaluated in adolescents only.
Occurrence of interruption or discontinuation of study drug(s) due to TEAE | Up to 5 Years
  A TEAE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Occurrence of laboratory abnormalities | Up to 5 Years
  As assessed by the NCI-CTCAE grading system (≥ Grade 3 or higher)
Concentrations of fianlimab in serum over time | Up to 5 Years
  The concentrations of fianlimab over time will be summarized by descriptive statistics by study arm for the overall population and for adolescent patients.
Concentrations of cemiplimab in serum over time | Up to 5 Years
  The concentrations of cemiplimab over time will be summarized by descriptive statistics by study arm for the overall population and for adolescent patients.
Concentration of finalimab anti-drug antibodies (ADA) and neutralizing antibodies | Up to 5 Years
  Immunogenicity will be characterized per drug molecule by ADA and NAb status.
Concentration of cemiplimab anti-drug antibodies (ADA) and neutralizing antibodies | Up to 5 Years
  Immunogenicity will be characterized per drug molecule by ADA and NAb status.
Patient report outcomes (PRO) for adults as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC-QLQ-C30) | Up to 5 Year
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. More points are considered to have a better outcome.
PRO for adults as measured by the European Quality of Life Dimension 5 (EQ-5D-5L) | Up to 5 Years
  The EQ-5D-5L a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
PRO for adults as measured by the Functional Assessment of Cancer Therapy (FACT) - melanoma | Up to 5 Years
  The FACT-M is a melanoma-specific quality of life questionnaire that is composed of items from the Functional Assessment of Cancer Therapy-General (FACT-G). The FACT-M is scored on a 5 point Likert-scale: "Not at all", "A little bit", "Somewhat", "Quite a bit", and "Very much.". A Higher score represents higher Health Related Quality of Life (HRQoL).
PRO for adults as determined by the Patient Global Impressions Scale (PGIS) | Up to 5 Years
  The PGIS is a single 1-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time by using a 4-point Likert scale that ranges from (1) = "none (no symptoms)" to (4) = "severe".
PRO for adults as determined by the Patient Global Impressions of Change Scale (PGIC) | Up to 5 Years
  The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change since starting treatment as rated on a 5-point Likert scale anchored by (1) "much better" to (5) "much worse", with (4) = "no change".
Time to global health status/quality of life deterioration per EORTC QLQ-C30 | Up to 5 years
Time to physical functioning deterioration per EORTC QLQ-C30 | Up to 5 Years
Time to role functioning deterioration per EORTC QLQ-C30 | Up to 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (211):
- United States (28):
  - UC San Diego, La Jolla, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - John Wayne Cancer Institute (JWCI), Santa Monica, California
  - The Melanoma And Skin Cancer Institute, Englewood, Colorado
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Orlando Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke Cancer Institute, University Hospital, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University James Comprehensive Cancer Center, Columbus, Ohio
  - St Lukes University Health Network, Easton, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Tennessee Oncology - Centennial Clinic Location, Nashville, Tennessee
  - Verdi Oncology, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
- Argentina (6):
  - Fundacion Centro de Investigaciones para la Transformacion (CENIT), Caba, Buenos Aires
  - Centro de Investigacion Pergamino, Pergamino, Buenos Aires
  - Clinica Viedma S.A., Viedma, Río Negro Province
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - DIABAID - Instituto de Asistencia Integral en Diabetes, Caba
- Australia (10):
  - Blacktown Cancer and Haematology Centre - Blacktown Hospital, Blacktown, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Liverpool Hospital - Cancer Therapy Centre, Liverpool, New South Wales
  - Melanoma Institute of Australia, Wollstonecraft, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Calvary North Adelaide Hospital, North Adelaide, South Australia
  - Eastern Health, Box Hill, Victoria
  - Andrew Love Cancer Centre, Geelong, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - One Clinical Research at Hollywood Private Hospital, Nedlands, Western Australia
- Belgium (3):
  - Vitaz campus Sint-Niklaas Moerland, Sint-Niklaas, Oost-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
- Brazil (18):
  - Hospital das Clinicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Liga Paranaense de Combate ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - INCA Instituto Nacional de Cancer, Santo Cristo, Rio de Janeiro
  - Oncosite Centro De Pesquisa Em Oncologia, Ijuí, Rio Grande do Sul
  - Instituto do Cancer em Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de vento, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia PUCRS, Porto Alegre, Rio Grande do Sul
  - Catarina Pesquisa Clinica, Itajaí, Santa Catarina
  - Instituto Joinvilense de Hematologia e Oncologia, Joinville, Santa Catarina
  - Animi Unidade de Tratamento Oncologico, Lages, Santa Catarina
  - Fundacao Pio XII - Hospital de Amor, Barretos, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto - Hospital de Base, São José do Rio Preto, São Paulo
  - Unimed Sorocaba, Sorocaba, São Paulo
  - Instituto COI, Rio de Janeiro
  - Hemomed, São Paulo
  - Hospital Sirio Libanes, São Paulo
  - Sao Camilo Oncologia, São Paulo
- Canada (4):
  - Dr. Everett Chalmers Hospital, Fredericton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Chile (3):
  - Oncocentro APYS, Viña del Mar, Región de Valparaíso
  - Clinica UC San Carlos de Apoquindo, Santiago, Santiago Metropolitan
  - Centro Oncologia de Precision Universidad Mayor, Santiago, Santiago Metropolitan
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno, Brno Mesto
  - University Hospital Hradec Kralove, Hradec Králové, North Central Czech Republic
  - University Hospital Ostrava, Ostrava
- France (21):
  - Centre Georges Francois Leclerc, Dijon, Bourgogne-Franche-Comté
  - CHU-Dijon, Dijon, Burgundy
  - Besancon Regional University Hospital Center, Besançon, Doubs
  - Chu De Bordeaux, Bordeaux, Gironde
  - Institut Claudius Regaud, IUCT-Oncopole, Toulouse, Haute-Garonne
  - CHU de Lille, Lille, Hauts-de-France
  - Service de Dermatologie CHU Saint Eloi, Montpellier, Herault
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche, Isere
  - Centre Francois Baclesse (CFB), Caen, Normandy
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - CHU Amiens-Picardie, Amiens, Picardie
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - N_Hôpital Ambroise-Paré, Boulogne-Billancourt
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire De Nice Hopital De L Archet, Nice
  - Centre Hospitalier de Valence, Valence
  - Institut Gustave Roussy, Villejuif
  - Hopital Avicenne, Bobigny, Île-de-France Region
  - Hospital Henri Mondor, Créteil, Île-de-France Region
  - Saint Louis Hospital, Paris, Île-de-France Region
- Georgia (7):
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi, Caucasus
  - Cancer Center of Adjara, Batumi
  - Acad.Fridon Todua Medical Center- Research Institute of Clinical Medicine, Tbilisi
  - Israeli Georgian Medical Research Clinic Helsicore, Tbilisi
  - LTD New Hospitals, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - TIM - Tbilisi Institute of Medicine, Tbilisi
- Germany (22):
  - University Medical Center Mannheim, Mannheim, Baden-Wurttemberg
  - University of Tuebingen, Tübingen, Baden-Wurttemberg
  - University Hospital Augsburg, Augsburg, Bavaria
  - Dermatology Erlangen, Erlangen, Bavaria
  - LMU Klinikum, Munich, Bavaria
  - University Hospital of Regensburg, Regensburg, Bavaria
  - Klinikum Darmstadt GmbH, Darmstadt, Hesse
  - University Clinic Frankfurt, Frankfurt am Main, Hesse
  - University Medical Center Goettingen, Göttingen, Lower Saxony
  - Helios Kliniken Schwerin, Schwerin, Mecklenburg-Vorpommern
  - Ruhr University Bochum, Bochum, North Rhine-Westphalia
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - University Hospital Muenster, Münster, North Rhine-Westphalia
  - Fachklinik Hornheide, Münster, North Rhine-Westphalia
  - Hautklinik, Ludwigshafen am Rhein, Rhineland-Palatinate
  - University Hospital Dresden, Dresden, Saxony
  - Skin Cancer Center Harz, Quedlinburg, Saxony-Anhalt
  - University Hospital of Universitatsklinikum Schleswig Holstein (UKSH) Campus Kiel, Kiel, Schleswig-Holstein
  - Universitatsklinikum Schleswig Holstein Campus Luebeck, Lübeck, Schleswig-Holstein
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - Charite Universitaetsmedizin Berlin, Berlin
  - Klinikum Bremen Ost, Bremen
- Greece (5):
  - National and Kapodistrian University of Athens, Athens, Attica
  - Metropolitan Hospital, Neo Faliro, Attica
  - Ongology Theageneio Thessaloniki, Thessaloniki
  - BioClinic Thessaloniki, Thessaloniki
  - Interbalkan Medical Center, Thessaloniki
- Ireland (4):
  - Galway University Hospital, Galway, Connacht
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St Vincents University Hospital, Dublin
- Israel (3):
  - Haemek Medical Center, Afula, Northern District
  - Hadassah Medical Organization, Jerusalem
  - Sheba Medical Center, Tel Litwinsky
- Italy (14):
  - Clinica Oncologica, AOU Riuniti Ancona, Ancona, An
  - U.O.C. Oncologia Medica ed Ematologia (U.O.C Medical Oncology and Hematology), Naples, Campania
  - Istituto Romagnolo per lo Studio dei Tumori (IRST), Meldola, Forli Cesena
  - Istituto Clinico Humanitas, Milan, Lombardy
  - Istituto dei Tumori, Bari
  - Azienda Ospedaliera Santa Croce i Carle, Cuneo
  - Istituto Europeo di Oncologia, Milan
  - Instituto Nazionale Tumori Fondazione Giovanni Pascale, Naples
  - University of Perugia, Perugia
  - Fondazione Policlinico Universitrio a. Gemelli - IRCCS, Rome
  - Campus Bio-Medico di Roma, Rome
  - Istituto Dermopatico dell'Immacolata, Rome
  - Santa Chiara Hospital, Trento
  - Azienda Sanitaria Universitaria del Friuli Centrale, Udine
- Mexico (7):
  - Preparaciones Oncologica SC, León, Guanajuato
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Pan American Clinical Research, Guadalajara, Jalisco
  - iCan Oncology, Monterrey, Nuevo León
  - Neurociencias Estudios Clinicos SC, Culiacán, Sinaloa
  - Centro De Atencion E Investigacion Clinica En Oncologia SCP, Mérida, Yucatán
  - Faicic Centro de Investigacion Clinica de Veracruz, Veracruz
- Poland (5):
  - Mazowiecki Szpital Wojewodzki, Siedleckie Centrum Onkologii, Siedlce, Mazxowieckie
  - UCK, Gdansk, Pomeranian Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o.Wojewodzie Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Słupsku Sp. z o.o., Słupsk, Pomeranian Voivodeship
  - Poznan University of Meidcla Science, Poznan, Wielkopolska
- Romania (8):
  - Institute of Oncology Bucharest, Bucharest, București
  - Cardiomed, Cluj-Napoca, Cluj
  - Institute of Oncology Prof. Dr Ion Chirircuta, Cluj-Napoca, Cluj
  - Radiotherapy Center Cluj, Floreşti, Cluj
  - Sfantul Nectarie Oncology Center, Craiova, Dolj
  - Oncocenter Oncologie Clinica S.R.L, Timișoara, Timiș County
  - Oncomed, Timișoara, Timiș County
  - Centrul De Oncologie Euroclinic, Iași
- South Africa (4):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Wilgers Oncology Centre, Pretoria, Gauteng
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Cape Town Oncology Trials, Kraaifontein, Western Cape
- Spain (16):
  - H. Germans Trias i Pujol, ICO-Badalona, Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Instituto Oncologico Dr Rosell Hospital Universitari Quiron Dexeus Location, Barcelona, Catalonia
  - Hospital Universitario Central De Asturias, Oviedo, Principality of Asturias
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Catalan Institute of Oncology (ICO) Hospitalet, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre Universidad Complutense de Madrid UCM, Madrid
  - Hospital Universitario La Pa<, Madrid
  - Centro Integral Oncologico HM Clara Campal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - Incliva - Instituto de Investigacion Sanitaria, Valencia
- Turkey (Türkiye) (11):
  - Baskent University, Yüreğir, Adana
  - Dicle University - Medical Faculty Campus, Sur, Diyarbakır
  - Kocaeli University, İzmit, Kocaeli
  - Gaziantep Medicalpoint Hospital, Gaziantep, Sehitkamil
  - Gulhane Research And Training Hospital, Ankara
  - Ozel Liv Hospital, Ankara
  - Sbu Doctor Abdurrahman Yurtaslan Ankara Onkoloji Suam, Ankara
  - Memorial Ankara Hospital, Ankara
  - Trakya University, Edirne
  - Istanbul University Cerrahpasa at Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Medeniyet University - Prof Dr Suleyman Yalcin Sehir Hospital, Istanbul
- United Kingdom (9):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Edinburgh Cancer Centre, Edinburgh, Lothian
  - Bristol Haematology And Oncology Centre (BHOC) - Bristol Cancer Institute, Bristol, Somerset
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University Hospital Coventry and Warwickshire Nhs Trust, Coventry, West Midlands
  - Saint Bartholomew's Hospital, London
  - University College London Hospitals, London
  - The Christie, Manchester
  - Taunton and Somerset NHS Foundation Trust, Taunton

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: A clinical study for adults and adolescents who are melanoma-free following surgery. — https://harmonyadjuvantmelanomastudy.com/